CLINICAL TRIAL: NCT05758571
Title: Oxygen Atomizing Inhalation of EGCG in the Treatment Interstitial Pneumonia in Cancer Patients: Phase I-II Clinical Trial
Brief Title: Oxygen Atomizing Inhalation of EGCG in the Treatment Interstitial Pneumonia in Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Han Xi Zhao, Principal investigator, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTEBC-2023
Record Dates: First submitted 2023-02-08; First posted 2023-03-07 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Interstitial Pneumonia; Neoplasms Malignant
Keywords: EGCG
MeSH Terms: conditions — Lung Diseases, Interstitial; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EGCG（Epigallocatechin-3-gallate ） (Experimental): Epigallocatechin-3-gallate (EGCG) (high pressure liquid chromatographic purity ≥ 95%; from Ningbo Hepu Biotechnology Co., Ltd.) is dissolved in 0.9% normal saline; 10ml is inhaled by atomization three times a day. From the beginning of the diagnosis and 7 days after the signing of the informed consent form, the medication can be continued according to the wishes of the patients, but the total medication time is not more than 14 days.
  Interventions: Drug: EGCG

INTERVENTIONS:
Drug: EGCG — EGCG (high pressure liquid chromatographic purity ≥ 95%; from Ningbo Hepu Biotechnology Co., Ltd.) is dissolved in 0.9% normal saline; 10ml is inhaled by atomization three times a day.
  Other Names: epigallocchin-3-gallate

SUMMARY:
Epigallocatechin-3-gallate (EGCG) is a major polyphenol of green tea that possesses a wide variety of actions, such as anti-inflammatory, anti-fibrotic, pro-apoptotic, anti-tumorous, and metabolic effects via modulation of a variety of intracellular signaling cascades. In addition, preclinical studies have also emphasized the antiviral activity of epigallocatechin-3-gallate (EGCG), including SARS-CoV-2.

In previous studies, we found that EGCG can prevent and cure radiation-induced normal tissue damage in tumor patients. In clinical studies, we found that EGCG can prevent and treat radiation-induced acute radiation esophagitis, acute radiation skin injury, acute radiation oral mucositis with high safety. Thus, we designed this phase I-II clinical study in order to investigate the possible role of EGCG in the treatment interstitial pneumonia in tumor patients.

DETAILED DESCRIPTION:
In this phase I study, subjects were divided into four dose groups according to the improved Fibonacci method and were given different doses of EGCG to evaluate adverse events. At the same time, the researchers conducted a phase II study of EGCG in tumor patients with interstitial pneumonia. The Phase II study was conducted with a randomized, controlled, placebo dose determined by Phase I. the subjects were divided into two groups (experimental group and placebo group). To observe the effectiveness of EGCG, the researchers will use both clinician assessment and patient self-assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed malignant tumors by pathology or cytology
* COVID-19 with a confirmed positive polymerase chain reaction or antigen test result for SARS-CoV-23
* Moderate pneumonia, according to the diagnosis and treatment standard of COVID-19 in Peking Union Medical College Hospital
* Pulmonary function of the patient can be treated with aerosol inhalation for 5-7 days

Exclusion Criteria:

* Current or recent progresses rapidly and may develop into a Critical illness with coronavirus in a short period of time
* Caused by other viruses such as cytomegalovirus, as well as pneumocystis pneumonia, pulmonary edema, aspiration pneumonia and acute interstitial pneumonia
* Any condition including medical, emotional, psychiatric, or logistical that, in the opinion of the Investigator would preclude the participant from adhering to the protocol or would increase the risk associated with study participation
* Need systemic use of immune suppressive agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With EGCG-Related Adverse Events as Assessed by CTCAE v4.0 | through study completion, an average of 1 year
  CTCAE v4.0 is an international standard for evaluating adverse event to cancer treatment.
Changes of imaging examination (chest CT) after administration | up to 2 weeks
  The changes of lung before and after treatment were judged by CT chest with or without contrast.

CONTACTS AND LOCATIONS:
Overall Officials: Ligang Xing, MD, PhD, Study Chair — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China

REFERENCES:
- [Derived] Yin X, Zhu W, Tang X, Yang G, Zhao X, Zhao K, Jiang L, Li X, Zhao H, Wang X, Yan Y, Xing L, Yu J, Meng X, Zhao H. Phase I/II clinical trial of efficacy and safety of EGCG oxygen nebulization inhalation in the treatment of COVID-19 pneumonia patients with cancer. BMC Cancer. 2024 Apr 17;24(1):486. doi: 10.1186/s12885-024-12228-3. PMID 38632501